CLINICAL TRIAL: NCT03142659
Title: Evaluation and Management of Heart Failure Patients
Status: Recruiting | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Eli Sprecher, MD, Head of Research and development, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-16-ML-0574-16-TLV-CTIL
Record Dates: First submitted 2017-05-01; First posted 2017-05-05 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: registry-no intervention — registry-no intervention After filling the informed consent the patients will be evaluated for clinical history and physical examination by the nurse and a cardiologist. Then, the patients may perform the following test: ECG, Chest X-RAY, Blood test including: complete blood count, renal and liver function, electrolytes, thyroid function, cholesterol, glucose, Troponin and Brain Natriuretic Peptide

SUMMARY:
The investigator is trying to improving our knowledge in the treatment of HF patients, for the purpose of improving their quality of life and reducing hospitalizations. For achieving this the investigator would like to build a registry which will include all the HF patients going an evaluation in the Heart Failure unit or clinic in our facility,

DETAILED DESCRIPTION:
The prevalence of Heart Failure depends on the definition applied, but is approximately 1-2% of the adult population in developed countries, rising to ≥10% among people >70 years of age. Among people >65 years of age presenting to primary care with breathlessness on exertion, one in six will have unrecognized HF. The lifetime risk of HF at age 55 years is 33% for men and 28% for women. The most recent European data (ESC-HF pilot study) demonstrate that 12-month all-cause mortality rates for hospitalized and stable/ambulatory HF patients were 17% and 7%, respectively, and the 12-month hospitalization rates were 44% and 32%, respectively. Modifying risk factors and dynamic change of the medical treatment may improve symptoms, quality of life and reduce hospitalization due to HF exacerbation. For this cause, the Heat Failure unit was established. The goal of the Heart Failure unit is to provide medical and nursing follow-up for severe HF patients with New York Heart Association Function III-IV in purpose to improve their quality of life and reduce hospitalizations. At each visit the patients will be evaluated by a nurse and a cardiologist, blood tests will be performed and IV treatment will be given as needed, including Furosemide, Iron, Dobutamine and Packed Cells.

The investigator is trying to improving our knowledge in the treatment of HF patients, for the purpose of improving their quality of life and reducing hospitalizations. For achieving this the investigator would like to build a registry which will include all the HF patients going an evaluation in the Heart Failure unit or clinic in our facility. Prospective registry which will include all the HF patients evaluated in the Heart Failure unit or clinic. The patients will sign an informed consent form. After filling the informed consent the patients will be evaluated for clinical history and physical examination by the nurse and a cardiologist. Then, the patients may perform the following test: ECG, Chest X-RAY, Blood test including: complete blood count, renal and liver function, electrolytes, thyroid function, cholesterol, glucose, Troponin and Brain Natriuretic Peptide. It is impotent to mentions that all of the test mentioned above are being performed as part as the Heart Failure unit treatment and none are being done for the purpose of the study. After completing the evaluation the patients will be treated as needed by IV medications such as Furosemide, Iron, Dobutamine and Packed Cells. The data collected will include demographic: gender, age, hospitalization, diagnosis, symptoms, clinical as well as laboratory, echocardiographic and echocardiogram findings.

Identified details will be separated in a way that will not enable to review them. All data handling and the separation of the identified data will be done by the Principal Investigator, or sub-investigator in this study, who is in charge of the hearing screening program in our institution.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Patient evaluated in the Heart Failure unit or clinic in our facility.
3. Approved consent.

Exclusion Criteria:

1. Patients who haven't signed the informed consent in the prospective group.

Ages: 18 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Prospective registry which will include all the HF patients evaluated in the Heart Failure unit or clinic and will sign an informed consent form
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
NP/ pro-BNP from baseline | 10 years
QT measurements | 10 years
  ECG will be performed at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Michal Laufer Perl, MD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel